CLINICAL TRIAL: NCT03023579
Title: The Star Excursion Balance Test: Analysis of Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Do hyun Kim, Principal Investigator, Inje University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DKim
Record Dates: First submitted 2017-01-11; First posted 2017-01-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Search MeSH

ARMS (1):
- The star excursion balance test (Experimental): The star excursion balance test: simple test for dynamic balance
  Interventions: Other: The star excursion balance test

INTERVENTIONS:
Other: The star excursion balance test

SUMMARY:
PURPOSE: The investigators estimated the reliability, standard error of measurement (SEM), and minimum detectable change (MDC) of the star excursion balance test (SEBT) in children with cerebral palsy (CP).

METHODS: Eight children with CP (four boys and four girls, sixteen legs) participated in this study. Each child carried out the SEBT and was assessed by two examiners. To determine intra-rater reliability, the investigators calculated the intra-class correlation coefficient (ICC) model (3,3). The investigators also calculated the ICC model (2,3) to determine the inter-rater reliability.

ELIGIBILITY:
Inclusion Criteria:

* were aged between 4 and 12 years,
* had a status above level II on the Gross Motor Function Classification System (GMFCS),
* were able to understand instructions from the rater, and

Exclusion Criteria:

* had history of fracture or sprain of the lower limbs over the previous 12 months.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The star excursion balance test | 6 months